CLINICAL TRIAL: NCT02245321
Title: Caring for Those Who Share: Mitigating Iron Deficiency In Regular Blood Donors
Brief Title: Strategies to Reduce Iron Deficiency
Acronym: STRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Westat (Other)
Collaborators: Versiti Blood Health (Other); American National Red Cross (Other); The Institute for Transfusion Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01HL10580901
Record Dates: First submitted 2014-09-10; First posted 2014-09-19 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Iron Deficiency
Keywords: hemoglobin recovery; iron recovery; iron supplements
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous gluconate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Letter Group- No information (Placebo Comparator): Receive a thank you letter after each blood donation.
  Interventions: Other: Letter - No Information Provided
- Letter Group- Information Provided (Experimental): Receive a letter informing them of their ferritin result at each visit, along with recommendations for blood donation.
  Interventions: Other: Letter Group- Information Provided
- Ferrous gluconate- 0 mg (Placebo Comparator): Receive pills to take daily that contain no iron (a placebo or inert pill).
  Interventions: Dietary Supplement: Placebo
- Ferrous gluconate- 19 mg (Experimental): Receive pills to take daily that contain 19 mg of iron (the typical amount in a multivitamin with iron).
  Interventions: Dietary Supplement: Ferrous gluconate- 19 mg
- Ferrous gluconate- 38 mg (Experimental): Receive pills to take daily that contain 38 mg iron (the typical amount in an over-the-counter iron supplement).
  Interventions: Dietary Supplement: Ferrous gluconate- 38 mg

INTERVENTIONS:
Dietary Supplement: Ferrous gluconate- 19 mg — Receive pills to take daily that contain 19 mg of iron (the typical amount in a multivitamin with iron).
  Arms: Ferrous gluconate- 19 mg
Dietary Supplement: Ferrous gluconate- 38 mg — Receive pills to take daily that contain 38 mg iron (the typical amount in an over-the-counter iron supplement).
  Arms: Ferrous gluconate- 38 mg
Other: Letter Group- Information Provided — Receive a letter informing them of their ferritin result at each visit, along with recommendations for blood donation.
  Arms: Letter Group- Information Provided
Other: Letter - No Information Provided — Receive a letter thanking the participant for their participation.
  Arms: Letter Group- No information
Dietary Supplement: Placebo — Receive pills to take daily that contain 0 mg iron.
  Arms: Ferrous gluconate- 0 mg

SUMMARY:
The prevalence of iron deficiency in blood donors has been demonstrated to be a direct consequence of repeat blood donations. Given the adverse effects of iron deficiency, it is priority to implement programs to remediate iron deficiency issues associated with blood donations. To explore this issue, the study's aims to:

1. Determine whether regular blood donors provided with accurate information about their iron status and written recommended courses of action will take steps to prevent/mitigate iron deficiency on their own without being given iron supplements by the blood center; and
2. Determine if two different amounts of iron provided by the blood center will prevent/mitigate iron deficiency in regular blood donors.

To conduct this randomized, placebo controlled study, participant donors will be assigned to one of two arms and followed for a 24 month period. Each subject will provide additional blood samples of 7 ml and 4.5 ml at each study visit for the purpose of tracking hemoglobin (Hgb), ferritin, soluble transferrin receptor (sTfR), and hematology laboratory results.

Under the two study arms, subjects are to be randomized into one of the following five blinded categories:

* Receive a thank you letter after each blood donation.
* Receive a letter informing them of their ferritin result at each visit, along with recommendations for blood donation.
* Receive pills to take daily that contain no iron (a placebo or inert pill).
* Receive pills to take daily that contain 19 mg of iron (the typical amount in a multivitamin with iron).
* Receive pills to take daily that contain 38 mg iron (the typical amount in an over-the-counter iron supplement).

DETAILED DESCRIPTION:
Inclusion Criteria

* Donors who have donated whole blood or double red cells ≥ 2 times in the last 12 months if female, or, ≥ 3 times in the last 12 months if male.
* Commitment to meet the donation frequency requirement for the study for two more years, give a blood sample at each visit, and complete baseline and follow-up surveys.

Exclusion Criteria

* Subjects < 18 years of age.
* Subjects taking iron supplements (including multivitamins with iron) up to one month prior to enrollment.
* Females who are pregnant or plan to become pregnant in the following 2 years.
* Subjects unwilling to meet the requirements of the study.

ELIGIBILITY:
Inclusion Criteria:

* Repeat donors who have previously participated in RISE study and have continued to donate at a required frequency (donated whole blood or double red cells ≥ 2 times in the last 12 months if female, or, ≥ 3 times in the last 12 months if male)
* Non-RISE donors who have donated whole blood or double red cells ≥ 2 times in the last 12 months if female, or, ≥ 3 times in the last 12 months if male
* commitment to meet the donation frequency requirement for this study for two more years, give a blood sample at each visit, and complete baseline and follow-up surveys

Exclusion Criteria:

* subjects < 18 years of age
* subjects taking iron supplements (including multivitamins with iron) up to one month prior to enrollment
* females who are pregnant or plan to become pregnant in the following 2 years
* subjects unwilling to meet the requirements of the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2011-06; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (HgB) | Change from baseline in HgB over 2 years
  a protein responsible for transporting oxygen in the blood

SECONDARY OUTCOMES:
Ferritin | Change from baseline in ferritin over 2 years
  a protein that stores iron and releases it when your body needs it
Soluble transferrin receptor (sTfR) | Change from baseline in sTfR over 2 years
  a protein receptor that is used as a measure of functional iron status and the investigation of iron deficiency anemia
Laboratory Hematology results | Change from baseline in Laboratory hematology results over 2 years.
  Hemoglobin, Hematocrit, Mean Corpuscular Value (MCV), Mean Corpuscular Hemoglobin (MCH)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Mast, MD, PhD, Principal Investigator — BloodCenters of Wisconsin
Locations (4):
- United States (4):
  - American Red Cross, Connecticut Region, Farmington, Connecticut
  - Westat, Rockville, Maryland
  - The Institute for Transfusion Medicince, Pittsburgh, Pennsylvania
  - BloodCenter of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Bialkowski W, Kiss JE, Wright DJ, Cable R, Birch R, D'Andrea P, Bryant BJ, Spencer BR, Mast AE. Estimates of total body iron indicate 19 mg and 38 mg oral iron are equivalent for the mitigation of iron deficiency in individuals experiencing repeated phlebotomy. Am J Hematol. 2017 Sep;92(9):851-857. doi: 10.1002/ajh.24784. Epub 2017 Jun 9. PMID 28494509
- [Result] Chansky MC, King MR, Bialkowski W, Bryant BJ, Kiss JE, D'Andrea P, Cable RG, Spencer BR, Mast AE. Qualitative assessment of pica experienced by frequent blood donors. Transfusion. 2017 Apr;57(4):946-951. doi: 10.1111/trf.13981. Epub 2017 Feb 5. PMID 28164344
- [Result] Mast AE, Bialkowski W, Bryant BJ, Wright DJ, Birch R, Kiss JE, D'Andrea P, Cable RG, Spencer BR. A randomized, blinded, placebo-controlled trial of education and iron supplementation for mitigation of iron deficiency in regular blood donors. Transfusion. 2016 Jun;56(6 Pt 2):1588-97. doi: 10.1111/trf.13469. Epub 2016 Jan 26. PMID 26813849
- [Result] Bialkowski W, Bryant BJ, Schlumpf KS, Wright DJ, Birch R, Kiss JE, D'Andrea P, Cable RG, Spencer BR, Vij V, Mast AE. The strategies to reduce iron deficiency in blood donors randomized trial: design, enrolment and early retention. Vox Sang. 2015 Feb;108(2):178-85. doi: 10.1111/vox.12210. Epub 2014 Dec 3. PMID 25469720